CLINICAL TRIAL: NCT03383302
Title: Stereotactic Body Radiotherapy Radiotherapy With Immunotherapy in Early Stage Non-small Cell Lung Cancer: Tolerability and Lung Effects
Brief Title: SBRT With Immunotherapy in Early Stage Non-small Cell Lung Cancer: Tolerability and Lung Effects
Acronym: STILE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4644
Record Dates: First submitted 2017-11-23; First posted 2017-12-26 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Non-small Cell Lung Cancer Stage II; Non-small Cell Lung Cancer Stage I
Keywords: Non-small cell lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Nivolumab

STUDY DESIGN:
Intervention Model Description: This is a single arm, phase Ib/II open label study of nivolumab administered on completion of SBRT to patients with early stage NSCLC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm 1 Tolerabilty (Experimental): This is a single arm study of nivolumab administered on completion of stereotactic body radiotherapy (SBRT) to patients with early stage NSCLC. The first 5 patients to enroll must have Eastern Co-operative Oncology Group (ECOG) performance status < 2 at the time of first dose of investigational medical product (IMP). An Independent Data Monitoring Committee (IDMC) will meet when the first 5 patients have reached 3 months follow up from their 1st dose of nivolumab or have withdrawn consent to follow-up. The IDMC, if satisfied with the safety data from the initial 5 patients, may recommend escalation to include recruitment of patients with ECOG performance status of 2.
  Interventions: Radiation: Stereotactic body radiotherapy; Drug: Nivolumab

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Patients will receive a total of 54 Gy if delivered in 3 fractions, 55 Gy if delivered in 5 fractions or 60 Gy if delivered in 8 fractions.
  Other Names: SBRT
Drug: Nivolumab — Nivolumab is a human immunoglobulin G4 (IgG4) monoclonal antibody, that binds to the PD-1 receptor and blocks interaction with its ligands PD-L1 and PD-L2. Nivolumab will be administered intravenously at a flat dose of 240 mg q2w over 30 minutes for 13 cycles followed by 480mg q4w over 60 minutes for 7 cycles, until 20 cycles in total to complete (a minimum of 1 year of treatment if no delays are encountered).
  Other Names: L01XC17; Opdivo

SUMMARY:
This is a single arm, multi-centre, phase II open label study of nivolumab with stereotactic body radiotherapy (SBRT) for early stage non-small cell lung cancer.

SBRT will be delivered in either 3 or 5 fractions for peripheral disease or 8 fractions in central disease. A flat dose of 240 mg nivolumab infusion will begin after the final fraction of SBRT, within 24 hours and typically on the same day. Nivolumab will subsequently be given every 2 weeks at a flat dose of 240 mg for a further 13 cycles followed by Nivolumab 480mg Q4W for 7 cycles until 20 cycles in total are complete, unless any study drug discontinuation criteria are met. Treatment (20 cycles) will take a minimum of 1 year to complete but may exceed this timeframe if treatment delays are encountered.

(Patients who have enrolled on Nivolumab Q2W 240mg regimen for 26 cycles and are beyond cycle 14 will receive 26 cycles Q2W in total to complete treatment).

Assessment of toxicities will be performed at each clinic visit during treatment, at 30 days after the final nivolumab infusion and until 100 days after the final nivolumab infusion. Changes in spirometry values and PFTs will be assessed throughout the trial.

Relapse rates will be assessed with staging CT scans at 3, 6, 12, 18 and 24 months post SBRT.

An exploratory assessment will be made of the effect pre-treatment pulmonary function tests (PFTs) have on outcome measures.

DETAILED DESCRIPTION:
This is a single arm, multi-centre, phase II open label study of nivolumab with stereotactic body radiotherapy (SBRT) for early stage non-small cell lung cancer.

Current United Kingdom (UK) guidelines for SBRT do not specify exclusion pulmonary function criteria. Severely reduced Forced Expiratory Volume in 1 second (FEV1) and diffusing capacity of the lung for carbon monoxide (DLCO) (<40% predicted) are common reasons for medical inoperability leading to the choice of SBRT. In a large prospective study of patients undergoing SBRT, poor baseline PFT was not predictive of toxicity including pneumonitis. At the 2 year follow up, the mean decline in percentage of predicted forced expiratory volume in one second (FEV1) and diffusion capacity of carbon monoxide (DLCO) were only 5.8% and 6.3% respectively. Focal SBRT is a well-tolerated procedure and acute complications are generally transient. Symptomatic radiation pneumonitis has been reported at rates of 4-25% of patients.

Drug induced pneumonitis is reported at 6% in lung cancer patients receiving nivolumab and at 2% with grade 3-4 toxicity. Of note, such rates are similar or lower to other drugs used in NSCLC including docetaxel for which no PFT restrictions occur. In this study, frequent assessment of spirometry values may help to predict patients that are developing subclinical pneumonitis and prompt for early intervention.

SBRT will be delivered in either 3 or 5 fractions for peripheral disease or 8 fractions in central disease. A flat dose of 240 mg nivolumab infusion will begin after the final fraction of SBRT, within 24 hours and typically on the same day. Nivolumab will subsequently be given every 2 weeks at a flat dose of 240 mg for a further 13 cycles followed by Nivolumab 480mg Q4W for 7 cycles until 20 cycles in total are complete, unless any study drug discontinuation criteria are met. The study will recruit 31 patients. We anticipate it will take approximately 18 months to recruit 31 patients.

The study will include subjects with histologically verified NSCLC deemed by a local multidisciplinary team (MDT) to have anatomical stage T1-3 [≤6cm] N0 M0 by means of computed tomography (CT) and fludeoxyglucose-positron emission tomography (FDG-PET) , amenable to radical treatment with SBRT and inoperable due to medical co-morbidity, being technically unresectable or patient declining surgery after offer of surgical assessment.

Subjects will receive nivolumab as per the treatment schedule unless any withdrawal criteria are met. The first nivolumab infusion will be given after the final fraction of SBRT, within 24 hours and generally on the same day. Clinical follow up and investigations are as detailed in the schedule of assessment.

The first 5 patients to enroll must have Eastern Co-operative Oncology Group (ECOG) performance status (PS) < 2 at the time of first dose of investigational medical product (IMP). An Independent Data Monitoring Committee (IDMC) will meet when the first 5 patients have reached 3 months follow up from their 1st dose of nivolumab or have withdrawn consent to follow-up. Patients that have enrolled but did not receive IMP will be replaced. The IDMC, if satisfied with the safety data from the initial 5 patients, may recommend escalation to include recruitment of patients with ECOG performance status of 2. Further patients of PS <2 may enroll while awaiting the outcome of the IDMC meeting.

The IDMC will perform a further safety review when the first 5 patients enrolled with ECOG performance status 2 have reached 3 months follow up from their final fraction of radiotherapy or have withdrawn consent to follow-up. Patients that have enrolled but did not receive IMP will be replaced. Further patients with ECOG performance status 2 will not be able to enroll unless recommendation is given by the IDMC. In the event that 5 PS 2 patients have not enrolled by the point that the 15th recruited patient has reached 3 months follow up, then there will be a further mandated IDMC meeting to assess safety data from the study. Patients may continue to enroll while awaiting the outcome of this IDMC meeting.

Assessment of toxicities will be performed at each clinic visit during treatment, at 30 days after the final nivolumab infusion and until 100 days after the final nivolumab infusion. Changes in spirometry values and PFTs will be assessed throughout the trial.

Relapse rates will be assessed with staging CT scans at 3, 6, 12, 18 and 24 months post SBRT.

An exploratory assessment will be made of the effect pre-treatment pulmonary function tests (PFTs) have on outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed and dated a Research Ethics Committee (REC) approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care
* Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory tests
* ECOG Performance status (PS) 0-2
* Minimum of first 5 patients to be PS 0-1
* PS 2 patients to be enrolled only following recommendation by the Independent Data Monitoring Committee (IDMC)
* Patients with histological diagnosis of NSCLC, all histological sub-types are eligible
* Not suitable for surgery because of medical co-morbidity, lesion is technically inoperable or patient declines surgery after surgical assessment (or option of assessment)
* Single or synchronous/metachronous primary NSCLC lesions, tumour stage T1-3 (≤6cm), N0 M0 (UICC v.8) as determined by the local MDT based on minimum investigations of CT chest/abdomen within 8 weeks and FDG-PET within 6 weeks of 1st fraction of SBRT. Where the radiological nodal status is equivocal then only eligible if possible nodal disease is subsequently confirmed as pathologically negative with mediastinoscopy or endoscopic bronchial or oesophageal ultra-sound biopsy as necessary
* For synchronous tumours one lesion must have a histological diagnosis of NSCLC. For the other lesion a radiological diagnosis of NSCLC as determined by lung MDT is sufficient. (Upon diagnosis of metachronous primary NSCLC these lesions require biopsy for trial entry)
* Metachronous (single) primary NSCLC lesions, tumour stage T1-3 (≤6cm) N0 M0 (UICC v.8) presenting after previous treatment of T1-3(≤6cm) N0 M0 (UICC v.8) with surgery or SBRT are eligible for inclusion. Lung constraints must be able to feasibly achieved (according to dose constraints in 7.1.2
* Tumour stage T1-3 termed as 'central' disease within 2cm of main airways and proximal bronchial tree, but not abutting these structures (ultra-central), are suitable for entry. Up to 5 patients with 'central' primary NSCLC (up to 2 lesions) can be enrolled and followed up for 3 months following their final fraction of radiotherapy at which stage an IDMC meeting is required to assess further 'central' primary NSCLC recruitment
* Screening laboratory values must meet the following criteria prior to commencement of treatment:

  i) WBCs ≥ 2000/μL ii) Neutrophils ≥1500/μL iii) Platelets ≥ 100 X10³/μL iv) Haemoglobin ≥ 9.0 g/dL v) Serum creatinine of ≤ 1.5 X ULN or creatinine clearance (CrCl)/glomerular filtration rate (GFR) > 40 mL/minute (using Cockcroft/Gault formula or as assessed by local practice)
  1. . Female CrCl= [(140- age in years) X weight in kg X 0.85) ÷ (72 X serum creatinine in mg/ dL)]
  2. . Male CrCl= [(140- age in years) X weight in kg X 1.00) ÷ (72 X serum creatinine in mg/ dL)] vi) AST ≤ 3 X ULN vii) ALT ≤ 3 X ULN viii) Total bilirubin ≤ 1.5 X ULN (except subjects with Gilbert Syndrome, who must have total bilirubin < 50 μmol/L)
* No prior adjuvant or foreseen neo-adjuvant or adjuvant chemotherapy is allowed
* Males and Females ≥ 18 years of age
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) in the screening period and within 24 hours prior to the start of study drug.
* Women must not be breastfeeding during the study treatment and for a period up to 23 weeks post treatment completion
* WOCBP must agree to follow instructions for method(s) of contraception during the study treatment and for a total of 23 weeks post treatment completion
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) for contraception for a total of 31 weeks post treatment completion.

Exclusion Criteria:

* Any tumour that is not clinically definable on the treatment planning CT scan e.g. surrounded by consolidation or atelectasis
* 'Ultra-central' tumours, i.e. those adjacent to the hilar structures, with the gross tumour volume directly abutting a main bronchus
* Subjects with active, known autoimmune disease. Subjects with Type I diabetes mellitus, residual hypothyroidism due to an autoimmune condition requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enrol.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of the first dose of study drug administration. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease
* Subjects with previous malignancies (except non-melanoma skin cancers, early stage NSCLC treated with SBRT or surgery and current lesion not considered to be relapsed NSCLC, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period
* Patient with known interstitial lung disease or active, non-infectious pneumonitis
* Previous conventional radiotherapy to the chest or mediastinum. Patients who have had previous breast radiotherapy may be eligible at the discretion of the Chief Investigator
* Any serious or uncontrolled medical disorder or active infection that, in the opinion of the Investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the subject to receive protocol therapy
* All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE v.4.0) or baseline before administration of study drug
* Subjects must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before the first dose of study treatment
* Subjects who received prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) or who have previously taken part in a randomized BMS clinical trial for nivolumab or ipilimumab
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Positive test for hepatitis B virus (HBV) using HBV surface antigen (HBVsAg) test or positive test for hepatitis C virus (HCV) using HCV ribonucleic acid (RNA) or HCV antibody test indicating acute or chronic infection

  o Patients with a positive HCV antibody but no detection of HCV RNA indicating no current infection are eligible
* Patients who have received a live vaccine within 30 days prior to the first dose of trial treatment
* History of allergy to study drug components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Assessment of lung toxicity (pneumonitis) from treatment with Nivolumab after SBRT for early stage NSCLC | Six months from final dose of SBRT administered for each patient
  Rate of grade ≥ 3 pneumonitis with nivolumab after stereotactic body radiotherapy (SBRT) within 6 months of the final fraction of SBRT. A rate that exceeds 20% will be deemed unacceptable and will lead to a rejection of the null hypothesis.

SECONDARY OUTCOMES:
Adverse events (toxicity) assessment using CTCAE v.4 | 24 months from last dose of SBRT
  Frequency of treatment related adverse events of all grades and grade ≥ 3 as per CTCAE v. 4 after treatment with Nivolumab following SBRT
Number of doses of Nivolumab received by patients within 16 weeks of commencing adjuvant nivolumab after SBRT for early stage NSCLC | Within 16 weeks of each patient commencing treatment with Nivolumab after SBRT
  The proportion of patients receiving at least 1, 2, 3, 4, 5 and 6 doses of Nivolumab within 16 weeks of commencing treatment with Nivolumab after SBRT for early stage NSCLC
Disease relapse | 24 months from last dose of SBRT
  To assess local, local-regional and distant disease relapse rates
Relapse at specified timepoints | 3, 6, 12 and 24 months from the date of first fraction of SBRT for each patient
  Local, loco-regional and distant rates of relapse at 3, 6, 12 and 24 months
Overall survival | Overall survival rate (OS) at 6, 12 and 24 months
  Overall survival rate (OS) of the 31 patients at 6, 12 and 24 months (and up to 5 years at 36, 48 and 60 months if data mature and available)
Disease free survival | Disease Free Survival (DFS) at 6, 12 and 24 months
  Disease Free Survival (DFS) rate of the 31 patients at 6, 12 and 24 months (and up to 5 years at 36, 48 and 60 months if data mature and available)
Health-related quality of life (HRQoL) using Patient Generated Subjective Global Assessment in patients treated with Nivolumab after SBRT for early stage NSCLC | 24 months from last dose of SBRT
  Estimation of HRQoL using the Patient Generated Subjective Global Assessment in patients treated with Nivolumab after SBRT for early stage NSCLC.
Health-related quality of life (HRQoL) using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) in patients treated with Nivolumab after SBRT for early stage NSCLC | 24 months from last dose of SBRT
  Estimation of HRQoL using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30).
HRQoL using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13) in patients treated with Nivolumab after SBRT for early stage NSCLC. | 24 months from last dose of SBRT
  Estimation of HRQoL in patients treated with Nivolumab after SBRT for early stage NSCLC using the Eurpoean Organisation for Research and Treatment of Cancer Ouality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13).

OTHER OUTCOMES:
Impact on lung function | 24 months from last dose of SBRT
  Assessment of rates of toxicity within percentage of predicted FEV1 bands & DLCO bands
OS rates in PD-L1 expressers (≥ 1%) and non-expressers (< 1%) | 24 months from last dose of SBRT
  OS rates at 6, 12 & 24 months will be described according to PD-L1 expression
DFS rates in PD-L1 expressers (≥ 1%) and non-expressers (< 1%) | 24 months from last dose of SBRT
  DFS at 6, 12 & 24 months will be described according to PD-L1 expression
OS rates (squamous and non-squamous) | 24 months from last dose of SBRT
  OS rates at 6, 12 & 24 months will be described according to squamous and non-squamous subgroups
DFS rates (squamous and non-squamous) | 24 months from last dose of SBRT
  DFS rates at 6, 12 & 24 months will be described according to squamous and non-squamous subgroups
Measuring immune cell responses with treatment | 4 years from recruitment of first patient
  Measuring change in T cell receptor sub-types during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Merina Ahmed, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: No